CLINICAL TRIAL: NCT02235311
Title: Optimal Dose of Proton Pump Inhibitors Following an Upper Gastrointestinal Bleed
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting and consenting participants
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1212917
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Upper Gastrointestinal Bleed
Keywords: Proton pump inhibitor; Upper gastrointestinal bleed; Ulcer healing
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pantoprazole twice daily (Active Comparator): Pantoprazole 40mg orally twice daily x 8 weeks after acute management of UGIB
  Interventions: Drug: Pantoprazole
- Pantoprazole once daily (Active Comparator): Pantoprazole 40mg orally once daily x 8 weeks after acute management of UGIB
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole 40mg orally daily x 8 weeks after acute management of UGIB
  Other Names: Protonix

SUMMARY:
Despite recommendations from clinical practice guidelines to discharge patients from the hospital on once daily proton pump inhibitors after acute management of UGIB, clinical practice is to use twice daily proton pump inhibitor therapy. The objective of this study will be to assess whether or not once daily pantoprazole is non-inferior to twice daily pantoprazole in ulcer healing with a dose of once daily versus twice daily proton-pump inhibitor following an upper gastrointestinal bleed. Additionally, this study will observe for any potential difference in safety for once daily versus twice daily proton pump inhibitors.

DETAILED DESCRIPTION:
There are few clinical practice guidelines for the management of a non-variceal, upper gastrointestinal bleed (UGIB). The 2012 guidelines released by the American College of Gastroenterology (ACG) indicate that for active bleeding or non-bleeding visible vessels or adherent clot, a bolus of 80 mg proton pump inhibitor followed by continuous infusion of 8 mg/hr infusion is to be used. Following 72 hours of infusion therapy, an oral proton pump inhibitor (PPI) may be used. If the clot is a flat pigmented spot or a clean ulcer base, an oral proton pump inhibitor may be used for management (without infusion) (Laine 2012). There are no recommendations made on once versus twice daily proton pump inhibitor. The 2010 American College of Physicians guideline recommends following the 72-hour infusion with once-daily proton pump inhibitors for duration as dictated by underlying etiology following upper gastrointestinal bleeding (UGIB) (Barkun 2012). This recommendation is graded 1C, with the decision to support once-daily over twice-daily dosing due to demonstrated effective ulcer healing for patients with peptic ulcer disease with once-daily dosing, and insufficient data to suggest twice-daily is superior to once-daily. There have been no head-to-head trials to evaluate once-daily versus twice-daily proton pump inhibitor following acute management of an endoscopic bleed. Additionally, studies suggest about 50% to 60% of proton pump inhibitors are being used without appropriate indications or at inappropriate dosages (Ali 2009).Safety concerns such as increased risk for Clostridium difficile infection , community acquired pneumonia, electrolyte abnormalities (hypomagnesemia), and fractures are becoming more prevalent warranting improved risk versus benefit examination of proton pump inhibitors including ascertainment of least effective dosing (Ali 2009, Sheen 2011). Despite recommendations to discharge patients after acute management of UGIB on once daily PPI therapy, clinical practice is to use twice daily proton pump inhibitor therapy. The objective of this study will be to examine if once daily pantoprazole is non-inferior to twice daily pantoprazole with regards to ulcer healing after acute management of an UGIB. In addition, because more evidence is emerging regarding safety concerns with proton pump inhibitors, the study will seek to examine if once daily versus twice daily therapy results in difference in safety or adverse reactions such as occurrence of rebleed, C. difficile diarrhea, or pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18 years and older; Upper GI bleed confirmed by endoscopy

Exclusion Criteria:

* Intensive Care Unit admission, Emergency endoscopic intervention required to control bleeding, Malignant appearing ulcers as determined by endoscopy, Previous documented treatment with twice daily PPI for other indication, Receiving twice daily PPI therapy prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08-17 (Actual); Study Completion 2015-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Ausmus, Pharm.D., Principal Investigator — University of Missouri-Health Care
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali T, Roberts DN, Tierney WM. Long-term safety concerns with proton pump inhibitors. Am J Med. 2009 Oct;122(10):896-903. doi: 10.1016/j.amjmed.2009.04.014. PMID 19786155
- [Background] Masso Gonzalez EL, Garcia Rodriguez LA. Proton pump inhibitors reduce the long-term risk of recurrent upper gastrointestinal bleeding: an observational study. Aliment Pharmacol Ther. 2008 Sep 1;28(5):629-37. doi: 10.1111/j.1365-2036.2008.03780.x. Epub 2008 Jun 26. PMID 18616644
- [Background] Holster IL, Kuipers EJ. Management of acute nonvariceal upper gastrointestinal bleeding: current policies and future perspectives. World J Gastroenterol. 2012 Mar 21;18(11):1202-7. doi: 10.3748/wjg.v18.i11.1202. PMID 22468083
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Barkun AN, Bardou M, Kuipers EJ, Sung J, Hunt RH, Martel M, Sinclair P; International Consensus Upper Gastrointestinal Bleeding Conference Group. International consensus recommendations on the management of patients with nonvariceal upper gastrointestinal bleeding. Ann Intern Med. 2010 Jan 19;152(2):101-13. doi: 10.7326/0003-4819-152-2-201001190-00009. PMID 20083829
- [Background] Sheen E, Triadafilopoulos G. Adverse effects of long-term proton pump inhibitor therapy. Dig Dis Sci. 2011 Apr;56(4):931-50. doi: 10.1007/s10620-010-1560-3. Epub 2011 Mar 2. PMID 21365243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants signed the consent form. One went on to complete the study; 1 was terminated by PI before starting the treatment and 1 was lost to follow-up before starting the treatment.
Period: Overall Study
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
Started | 1 | 2
Completed | 1 | 0
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Count of Participants; unit: Participants]
  Age >18 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
Weight [Median (Inter-Quartile Range); unit: kg] | 140 [140 to 140] |  | 140 [140 to 140]
Glasgow-Blatchford Score [Mean (Standard Deviation); unit: summary score] — Summary score of presenting symptoms ranging from 0 - 29 to assess the likelihood that a patient with an acute upper gastrointestinal bleeding will need to have medical intervention. Score of >6 associated with higher risk of needing intervention.
  summary score | 17 (NA) — Standard Deviation not calculable from one data value. |  | 17 (NA) — Standard Deviation not calculable from one data value.
Heart rate [Mean (Standard Deviation); unit: bpm] | 105 (NA) — Standard Deviation not calculable form one data value. |  | 105 (NA) — Standard Deviation not calculable form one data value.
Participants with orthostasis [Number; unit: participants] — Orthostasis is a decrease in blood pressure that happens soon after standing. Measured by taking blood pressure while seated and then on standing.
  participants | 0 |  | 0
Mean arterial pressure (MAP) [Mean (Standard Deviation); unit: mm Hg] | 76 (NA) — Standard Deviation not calculable from one data value. |  | 76 (NA) — Standard Deviation not calculable from one data value.
Platelets [Mean (Standard Deviation); unit: Platelets/mm^3] | 299 (NA) — Standard Deviation not calculable from one data value. |  | 299 (NA) — Standard Deviation not calculable from one data value.
Blood urea nitrogen (BUN) [Mean (Standard Deviation); unit: mg/dl] | 25 (NA) — Standard Deviation not calculable from one data value. |  | 25 (NA) — Standard Deviation not calculable from one data value.
Serum creatinine (SCr) [Mean (Standard Deviation); unit: mg/dL] | 0.7 (NA) — Standard Deviation not calculable from one data value. |  | 0.7 (NA) — Standard Deviation not calculable from one data value.
Positive fecal occult blood test (FOBT) [Count of Participants; unit: Participants] | 0 |  | 0
H. pylori (serum) positive [Count of Participants; unit: Participants] | 0 | 0 | 0
Appearance of ulcer (clean-based) [Count of Participants; unit: Participants] | 1 |  | 1
Appearance of ulcer (oozing, bleeding) [Count of Participants; unit: Participants] | 0 |  | 0
Melena present [Count of Participants; unit: Participants] | 1 |  | 1
Hematemesis present [Count of Participants; unit: Participants] | 1 |  | 1
Syncope [Count of Participants; unit: Participants] | 0 |  | 0
Hepatic disease [Count of Participants; unit: Participants] | 0 |  | 0
NSAID use [Count of Participants; unit: Participants] | 1 |  | 1
Warfarin use [Count of Participants; unit: Participants] | 0 |  | 0
Steroid use [Count of Participants; unit: Participants] | 0 |  | 0
Novel oral anticoagulant (NOAC) use [Count of Participants; unit: Participants] | 0 |  | 0
smoker [Count of Participants; unit: Participants] | 0 |  | 0
alcoholism [Count of Participants; unit: Participants] | 0 |  | 0
history of ulcers [Count of Participants; unit: Participants] | 0 |  | 0
history of bleed [Count of Participants; unit: Participants] | 0 |  | 0
endoscopic intervention required [Count of Participants; unit: Participants] | 0 |  | 0
transfusion required [Count of Participants; unit: Participants] | 0 |  | 0
Malignant cause identified [Count of Participants; unit: Participants] | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Ulcer Healing
Description: as defined by follow-up endoscopy per gastroenterology service, 8 weeks after UGIB acute management
Time Frame: 8 weeks
Population: 1 ulcer located in duodenum, clean-base; randomized single-blinded to proton pump inhibitor (PPI) twice daily
Measure: Count of Participants; unit: Participants
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Secondary Outcome: Rate of Rebleed
Description: Per patient report or as defined by follow-up endoscopy per gastroenterology service, 8 weeks after UGIB acute management
  High clinical suspicion of rebleed includes melena, hematochezia, confirmed by repeat endoscopy, requiring additional management
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

3. Secondary Outcome: Clostridium Difficile Diarrhea
Description: Clostridium difficile confirmed by polymerase chain reaction (PCR)
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

4. Secondary Outcome: Community-Acquired Pneumonia
Description: As defined by clinical suspicion and/or positive sputum culture requiring antibiotic treatment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks after randomization
Description: no adverse events collected for the Pantoprazole Once Daily Arm/Group
Arm/Group | Pantoprazole Twice Daily | Pantoprazole Once Daily
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
trial eliminated due to very low enrollment Poorly adopted by GI department due to fears of using once daily PPI despite available evidence Need for expansion to more sites for better enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No